CLINICAL TRIAL: NCT03551457
Title: Potential Therapeutic Response In Urogenital Tumors: Ex-Ovo Avian Embryo Patient Avatar
Brief Title: Potential Therapeutic Response In Urogenital Tumors
Acronym: Avatar
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Leonardo Oliveira Reis, Researcher MD, MSc, PhD, University of Campinas, Brazil
Other Study IDs: AVATAR
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Urogenital Neoplasms; Drug Therapy
Keywords: Patient Derived Xenograft; Treatment Response Phenotype; Personalised
MeSH Terms: conditions — Urogenital Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Biopsy — Patient-derived xenograft treatment response phenotype.

SUMMARY:
Preclinical models of urogenital carcinoma have been emerging as a way to pre-determine drug resistance before therapy is targeted. The implantation of tumor specimens in the chorioallantoic membrane (CAM) of the chicken embryo results in a high-efficiency graft, thus allowing large-scale studies of "tumor avatar". The aim of the study is to develop a tumor culture platform for treatment evaluation. Biopsies will be collected from primary tumors of patients and grafted onto the chorioallantoic membrane of chicken embryos. After tumor implantation at the CAM, tumor growth will be accompanied by imaging that will quantify tumor vascularization, tumor volume, and tumor blood flow. Following tumor growth, "avatars" will be divided into different treatments. Using the "tumor avatar" model together with patient tumors, the investigators will be able to observe the individualized tumor response for each patient in a treatment context, as well as determine the potential drug to be used in each case. These results may support a phenotype-based reading within 7-10 days.

DETAILED DESCRIPTION:
Introduction

1. Phenotypic Evaluation Model

   In 1874, William Roberts and John Tyndall observed the inhibition of cell growth on the agar plate. In the 1940s, Heatley suggested the use of filter paper discs containing antimicrobial solutions and introduced the "radial disc method".

   WHO released a report on the methodology and the reference method in 1975, which support the international standard of Clinical Laboratory Standards. The phenotype response of microorganisms to antibiotic treatment, comparing the proliferation of colonies might offer a rationale to the herein proposed tumor treatment response phenotype platform (patient-derived tumor avatar).
2. Cancer Treatment on Patient-Derived Xenografts (PDX)

   To propose an individualized treatment, it is necessary to know the tumor treatment response phenotype, which varies with the host. Studies using xenografts are being used to predict a response to certain drugs.
3. Chorioallantoic Membrane

The chorioallantoic membrane (CAM) assay has been used as a fast, reproducible method for antitumor drug testing in vivo. This assay has been widely used for the study of angiogenesis and has also been successfully developed in a xenograft tumor model, including urogenital tumors, due to the total non-development of the lymphoid system of the embryo. The new techniques have been studied, generating consequently new protocols. The major challenge for the xenograft model in CAM is a relatively high occurrence of embryonic death after egg removal, with a mortality rate between 25 and 50%.

The chick eggs will be used because they present a favorable vascularization environment. After the growth of the CAM, which is after 8 days of egg fertilization, access to the blood vessels is highly facilitated, causing them to be manipulated and observed. This makes it able to sustain systems and cells in the way that complex cancer studies can be done.

Blood vessels in addition to nourishing the development of -allo and xenografts, this redefined a supportive environment unique to intravasation and dissemination of tumor cells.

The CAM is highly vascularized, which makes it a rich medium for tumor implantation, in addition to other factors such as proteins. This support ends up being exclusive to the invasion, dissemination, and vascularization of tumor cells.

Treatment of genitourinary tumors is not yet individualized, due to the high heterogeneity of the tumors. The choice of treatment that the patient will get is defined by population studies that present inadequacies when transferred to the context of the individualized treatment.

The cell culture and organoids are a simple model to be applied, having a low cost and fast results. However, when the method is applied to the study of tumors, the results do not represent tumor environment conditions, forcing the cells to an adaptation that interferes with their growth and response to treatments patterns. Thus the xenografts models overcome some restrictions of the culture so that the framework is solid for its development. In contrast, the creation of a xenografts protocol becomes more complex, but it is a more representative method of cancer in its natural environment. CAM was studied with two strands, in-ovo, and ex-ovo. For in-ovo studies, the protocol was exposed by cutting eggshell.

The ex-ovo studies focus on improving the accessibility of the CAM and the embryo, enabling its documentation and manipulation.

Recently it has been described a correlation between renal tumors and drug resistance using exogenous CAM xenograft model. This causes other aspects to be monitored, studied and improved, especially regarding angiogenesis and research with tumors.

Hypothesis

There is increasing evidence that the diversity of the patient and cancer represent the main challenge in their treatment, which justifies the search for a clinical tool capable of providing information on the phenotype of response to treatment using the chorioallantoic tumor (CTA) platform/avatar.

Just as the antibiogram already established in clinical practice anticipates the susceptibility of bacteria to antibiotics, there is room for individualized treatment with potential benefit in cancer outcomes, quality of life and cost-effectiveness.

To define and anticipate the best treatment ("tumor chemogram") for each patient with urogenital cancer using treatment response phenotype platform, as the tumor avatar in the chorioallantoic membrane can transform the clinical practice.

Objectives

* To verify the efficiency of the sowing of fresh (immediate) and frozen tissue -80 degrees (in 24 and 48h) as a strategy in cases of failure of primary sowing;
* To evaluate the stability of the neoplastic tissue and the maintenance of its characteristics (genomic, proteomic, metabolic and phenotypic) in the proposed platform;
* To evaluate the response phenotype to the treatment of urogenital carcinomas in xenograft.
* To explore the impact of the proposed platform implementation on individualized treatment, its cost and results (oncological and functional) in patients with urogenital carcinomas.

Proposed Methodology

A prospective observational study including 30 biopsies of urogenital tumors from patients of the respective hospitals. Each biopsy will generate up to 12 tumor explants of 1 to 2 mm2, which will be implanted individually on the chorioallantoic membrane of 1 chicken embryo to test the 10 proposed drugs, plus 2 control eggs.

Therefore, 12 embryos will be needed for each biopsy. Biopsies of urogenital primary tumors of patients after consent will be collected, provided by the "Hospital das Clínicas da Unicamp" and "Hospital Municipal de Paulínia".

The material will be collected and placed in culture medium (McCoy) and kept on ice within 24 hours after resection. Part of the tissue fragments will be rapidly frozen and stored at -80oC for further studies.

It will be reserved a safety sample in ideal conditions of refrigeration for a sowing of rescue in cases of failure of the previous attempt. Samples will be divided where possible in:

* Fresh tumor: mitochondrial assay, culture, western blot
* Tumor formol: histopathology, immunohistochemistry
* Tumor culture: chorioallantoic membrane, frozen For the tumor biopsy graft, the CAM will be used when the embryos are 8 to 10 days old.

First, the CAM layer will be gently ruptured with the aid of a forceps, then the biopsy of the tumor will be placed near a Y-shaped bifurcation of a blood vessel. After placement of the tumor, 200ul of PBS will be placed to prevent contamination. After the graft comes into contact with the vascularization of the CAM, tumor growth will be monitored in a period of 3 to 4 days.

This process will be evaluated and if there is tumor growth the system will go to the treatment phase. Since there was tumor growth, the treatments will be performed from 17 days after the embryo. The treatments used will be doses of the following medicines: cisplatin, gemcitabine, paclitaxel, doxorubicin, carboplatin, pazopanib, sunitinib, sorafenib, methotrexate, and vinblastine. For the concentration of the drugs, they will be placed next to the filter paper in the tumor regions. This treatment will take from 3 to 4 days, after which analyzes will be carried out to determine the potentiality of each drug.

Euthanasia of the embryo will occur by decapitation (according to the protocol approved CEUA 4874-1 / 2018) since it already has a developed pain system.

Scissor cut through the CAM around the attached graft, transferred to a Petri dish with PBS. The excess of CAM will then be removed, leaving only the graft to be analyzed by histopathology, immunohistochemistry, western blotting and mitochondrial evaluation.

Risks

The risks involved in the participation of this study are minimal, as there is no interference in the treatment of the subject of the research, only the use of a small part of material withdrawn in the surgery that will be filed to be used in the laboratory in order to know even more about the disease, specifically identify future treatments with the best chances of results if necessary.

Benefits

This study will allow a greater knowledge of the disease with a potential benefit in the choice of future treatments, without altering any aspect of the current treatment that the research subject is receiving (the best standard treatment available at the time).

Data Analysis Methodology

Comparisons between primary tumor groups versus cultivated in xenograft will be performed using one-way ANOVA with the post hoc Bonferroni test. Data will be analyzed using Student t-tests or ANOVA repeated measures (Bonferroni post hoc test). The level of significance will be defined as less than 0.05 using Prism 5 (GraphPad software).

Primary outcomes

* Platform efficiency (tumor take in percentage)
* Platform representativeness (similarity between fresh and cultivated tumor)

Secondary outcomes

* Definition of tumor response phenotype to different therapeutic options.
* Impact of the proposed platform implementation on individualized treatment, its cost and results (oncological and functional)

ELIGIBILITY:
Inclusion Criteria:

* Urogenital neoplasm
* Undergo biopsy

Exclusion Criteria:

* Not accept to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 patients diagnosed with urogenital neoplasms, submitted to tumor ressection.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
- Therapeutic tumor response phenotype | 7 days
  drug sensitivity

SECONDARY OUTCOMES:
- Platform efficiency | 7 days
  tumor take in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo O Reis, MD, MSc, PhD, Principal Investigator — University of Campinas
Locations (1):
- Hospital das Clínicas Unicamp, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: End of study when data are published.
Access Criteria: Results shared in a publication.

REFERENCES:
- [Background] Chia S, Low JL, Zhang X, Kwang XL, Chong FT, Sharma A, Bertrand D, Toh SY, Leong HS, Thangavelu MT, Hwang JSG, Lim KH, Skanthakumar T, Tan HK, Su Y, Hui Choo S, Hentze H, Tan IBH, Lezhava A, Tan P, Tan DSW, Periyasamy G, Koh JLY, Gopalakrishna Iyer N, DasGupta R. Phenotype-driven precision oncology as a guide for clinical decisions one patient at a time. Nat Commun. 2017 Sep 5;8(1):435. doi: 10.1038/s41467-017-00451-5. PMID 28874669
- [Background] Dohle DS, Pasa SD, Gustmann S, Laub M, Wissler JH, Jennissen HP, Dunker N. Chick ex ovo culture and ex ovo CAM assay: how it really works. J Vis Exp. 2009 Nov 30;(33):1620. doi: 10.3791/1620. PMID 19949373
- [Background] Gao H, Korn JM, Ferretti S, Monahan JE, Wang Y, Singh M, Zhang C, Schnell C, Yang G, Zhang Y, Balbin OA, Barbe S, Cai H, Casey F, Chatterjee S, Chiang DY, Chuai S, Cogan SM, Collins SD, Dammassa E, Ebel N, Embry M, Green J, Kauffmann A, Kowal C, Leary RJ, Lehar J, Liang Y, Loo A, Lorenzana E, Robert McDonald E 3rd, McLaughlin ME, Merkin J, Meyer R, Naylor TL, Patawaran M, Reddy A, Roelli C, Ruddy DA, Salangsang F, Santacroce F, Singh AP, Tang Y, Tinetto W, Tobler S, Velazquez R, Venkatesan K, Von Arx F, Wang HQ, Wang Z, Wiesmann M, Wyss D, Xu F, Bitter H, Atadja P, Lees E, Hofmann F, Li E, Keen N, Cozens R, Jensen MR, Pryer NK, Williams JA, Sellers WR. High-throughput screening using patient-derived tumor xenografts to predict clinical trial drug response. Nat Med. 2015 Nov;21(11):1318-25. doi: 10.1038/nm.3954. Epub 2015 Oct 19. PMID 26479923
- [Background] Cully M. Cancer: Xenograft encyclopaedia identifies drug combination opportunities. Nat Rev Drug Discov. 2015 Dec;14(12):818. doi: 10.1038/nrd4788. Epub 2015 Nov 20. No abstract available. PMID 26585532
- [Background] Hagedorn M, Javerzat S, Gilges D, Meyre A, de Lafarge B, Eichmann A, Bikfalvi A. Accessing key steps of human tumor progression in vivo by using an avian embryo model. Proc Natl Acad Sci U S A. 2005 Feb 1;102(5):1643-8. doi: 10.1073/pnas.0408622102. Epub 2005 Jan 21. PMID 15665100
- [Background] Izumchenko E, Paz K, Ciznadija D, Sloma I, Katz A, Vasquez-Dunddel D, Ben-Zvi I, Stebbing J, McGuire W, Harris W, Maki R, Gaya A, Bedi A, Zacharoulis S, Ravi R, Wexler LH, Hoque MO, Rodriguez-Galindo C, Pass H, Peled N, Davies A, Morris R, Hidalgo M, Sidransky D. Patient-derived xenografts effectively capture responses to oncology therapy in a heterogeneous cohort of patients with solid tumors. Ann Oncol. 2017 Oct 1;28(10):2595-2605. doi: 10.1093/annonc/mdx416. PMID 28945830
- [Background] Skowron MA, Sathe A, Romano A, Hoffmann MJ, Schulz WA, van Koeveringe GA, Albers P, Nawroth R, Niegisch G. Applying the chicken embryo chorioallantoic membrane assay to study treatment approaches in urothelial carcinoma. Urol Oncol. 2017 Sep;35(9):544.e11-544.e23. doi: 10.1016/j.urolonc.2017.05.003. Epub 2017 May 25. PMID 28551413